CLINICAL TRIAL: NCT02930616
Title: A Comparison of pCLE Based Targeted Biopsy and WLE Based Standard Biopsy in Staging the Operative Link on Gastric Intestinal Metaplasia (OLGIM): A Randomized，Cross-over Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016SDU-QILU-17
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Intestinal Metaplasia; Confocal Laser Endomicroscopy; Operative Link on Gastric Intestinal Metaplasia; Biopsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Experimental): Patients in Group 1 will receive probe-based confocal endomicroscopy (pCLE) at first and Wight light endoscopy (WLE) 2 months later
  Interventions: Device: Patients in Group 1 will receive pCLE at first and WLE 2 months later
- goup 2 (Active Comparator): patients in Group 2 will receive WLE at first and pCLE 2 months later.
  Interventions: Device: patients in Group 2 will receive WLE at first and pCLE 2 months later.

INTERVENTIONS:
Device: Patients in Group 1 will receive pCLE at first and WLE 2 months later
  Arms: group 1
Device: patients in Group 2 will receive WLE at first and pCLE 2 months later.
  Arms: goup 2

SUMMARY:
Gastric intestinal metaplasia (GIM) is an important premalignant lesion for gastric cancer. Precisely surveillance of patients with GIM may result in early detection and improved prognosis. Though important, it is not necessary to recommend surveillance endoscopy for all patients with GIM, since the progression rate to gastric cancer within 10 years is only 1.8% in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older with Helicobacter pylori infection;
* Histologically verified GIM, atrophic gastritis or dysplasia.

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Conditions unsuitable for performance of pCLE, such as coagulopathy, impaired renal function or allergy to fluorescein sodium;
* Pregnancy or breastfeeding;
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the detection rate of each OLGIM (the Operative Link on Gastric Intestinal Metaplasia) stage by pCLE. | 9 months
the detection rate of each OLGIM (the Operative Link on Gastric Intestinal Metaplasia) stage by WLE. | 9 months

SECONDARY OUTCOMES:
the overall detection rate of GIM by pCLE. | 9 months
the overall detection rate of GIM by WLE. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No